CLINICAL TRIAL: NCT02374515
Title: Endocuff-assisted Colonoscopy: a Randomized Back-to-back Colonoscopy Study of Adenoma Detection.
Brief Title: Safety and Efficacy of Endocuff-assisted Colonoscopy for Adenoma Detection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Naples (Other)
Responsible Party: Principal Investigator, Giovanni Domenico De Palma, Full Professor of Surgery, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 230/14
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Adenomatous Polyps
MeSH Terms: conditions — Adenomatous Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endocuff assisted Colonoscopy (Active Comparator): Endocuff assisted Colonoscopy
  Interventions: Device: EndoCuff-assisted colonoscopy
- Standard Colonoscopy (Active Comparator): Standard colonoscopy
  Interventions: Device: Standard Colonoscopy

INTERVENTIONS:
Device: EndoCuff-assisted colonoscopy — Adenoma detection rate
  Other Names: EC-assisted colonoscopy
  Arms: Endocuff assisted Colonoscopy
Device: Standard Colonoscopy
  Arms: Standard Colonoscopy

SUMMARY:
This study investigated the impact of Endocuff-assisted colonoscopy on the adenoma detection rate at colonoscopy. This study involved patients undergoing elective screening or surveillance colonoscopy.

Patients were randomized to undergo Endocuff or regular, high-definition colonoscopy before undergoing a second colonoscopy by the alternate method. The primary outcome measure was the detection rate for adenomas between patients who underwent Endocuff first and patients who underwent regular colonoscopy first.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopy: Screening , Surveillance, Diagnostic

Exclusion Criteria:

* Pregnancy
* age<18 years
* age > 80 years
* known colonic strictures
* chronic inflammatory bowel disease
* active inflammation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate | 20 min.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni D. De Palma, MD, Principal Investigator — Federico II University
Locations (1):
- University of Naples Federico II, Naples, Italy